CLINICAL TRIAL: NCT01084382
Title: " Arthrospira Platensis" as Nutrition Supplementation for Female Adult Patients Infected by HIV in Yaoundé Cameroon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frank Winter (Other)
Collaborators: Centre Pasteur du Cameroun (Other)
Responsible Party: Sponsor-Investigator, Frank Winter, Dr., University of Giessen
Organization: University of Giessen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: JLU-AGKrawi_Spiru
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: HIV
Keywords: Arthrospira platensis; female HIV patient; Yaounde; Redox potential; Life quality; female patient infected by HIV in Yaounde: Cameroon
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthrospira platensis supplement (Active Comparator)
  Interventions: Dietary Supplement: Arthrospira platensis
- Protein/Dextran supplemented (Placebo Comparator)
  Interventions: Dietary Supplement: Arthrospira platensis

INTERVENTIONS:
Dietary Supplement: Arthrospira platensis — Patient take 5 gram supplement per day for 12 weeks in the first phase. In the second phase the two groups receive 5 gram per day of Arthrospira platensis for 12 weeks.
  One group will so haved received Arthrospira platensis for 24 weeks.
  Other Names: Group with supp.A; Group with supp.B,; for the first phase; in the second all patients receive supp.C

SUMMARY:
Early interests in Arthrospira p. (Spirulina) were based on its high source of protein. Recently, it has drawn attention for its therapeutic effects including anticancer properties, antiviral and antibacterial properties as well as improvement of the immune system.

The aim of this study is to investigate the effect of a daily supplementation with Spirulina for adult wife living with HIV/AIDS in Yaoundé.

DETAILED DESCRIPTION:
Several studies suggest that the micronutrient status determines the progression of the HIV infection to AIDS. This phenomenon may be explained by a vicious cycle of malnutrition and infection. Here, the immune system needs energy and micronutrients to adequately respond to infection. Early interests in Arthrospira p. (Spirulina) were based on its high source of protein. Recently, it has drawn attention for its therapeutic effects including reduction of blood cholesterol, nephrotoxicity, anticancer properties, radiation protection, antiviral and antibacterial properties as well here improvement of the immune system.

The aim of the three months Randomized, double blind and placebo Controlled Trial (RCT) is to investigate the effect of a daily supplementation with Spirulina for adult wife living with HIV/AIDS in Yaoundé. The trial will be experimental, prospective, and longitudinal on 70 patients. The study consists of two periods of three months.

The primary objective is to evaluate the efficacy of Spirulina on CD4+ T-lymphocyte count and the viral load during the RCT. The second objective is to confirm the effect of Spirulina on nutritional status markers: albumin, iron anemia, bioimpendenz, and BMI. The documentation of the nutritional marker will depict the restorative potential of Spirulina on patients with advanced HIV infection. Further data collected within a 24-hour recall will inform about the Individual Dietary Diversity Score. Explorative objective is the following of three disease outcomes of an HIV infection at four different time points, at t=0, 3, 6 months, and 1 month after the trial. The three explorative outcomes are the immune status with CD3+, CD8+, CD38+ and IFN gamma, the oxidative status, and the patient's quality of life.

This trial will end by August 2010.

ELIGIBILITY:
Inclusion Criteria:

* confirm Infection with HIV
* aged≥ 18-49 years
* BMI< 23

Exclusion Criteria:

* male
* under HAART
* pregnancy
* severe opportunistic infection requiring intensive medical care
* active smoking
* initiation of antioxidant vitamin therapy
* hyperlipidemia
* diabetes
* kidney/liver dysfunction
* intractable diarrhea (at least six liquid stools daily)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06-10 (Actual); Study Completion 2010-09-10 (Actual)

PRIMARY OUTCOMES:
CD4 cell account | 12 weeks

SECONDARY OUTCOMES:
Individual Dietary Diversity Score (IDDS) | 12-24 weeks
Quality of life perception (WHOQOL-HIV) | 12-24 weeks
immune status (CD3+, CD8+, CD38+ and IFN gamma) | 12-24 wekks
Anthropometric measurements (BMI, Bioimpedenz) | 12-24 weeks
Plasma redox potential (MDA,TAOS) | 12-24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Cameroon (2):
  - Hopital du jours, Yaoundé, Centre Region
  - "Hôpital du jours" from the Central Hospital, Yaoundé